CLINICAL TRIAL: NCT00639249
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Dose, Phase IIa Study of Safety and Motor Function Restoration in Subjects Treated With SA4503 Following Acute Ischemic Stroke
Brief Title: Safety and Preliminary Efficacy Study of SA4503 in Subjects Recovering From Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M's Science Corporation (Industry)
Responsible Party: Kazumasa Takao, M's Science Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ME1-2; EudraCT number: 2007-004840-60
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- P (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- A1 (Experimental): SA4503
  Interventions: Drug: SA4503 Low
- A2 (Experimental): SA4503
  Interventions: Drug: SA4503 High

INTERVENTIONS:
Drug: placebo — Oral administration
  Arms: P
Drug: SA4503 Low — Oral administration
  Arms: A1
Drug: SA4503 High — Oral administration
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of SA4503 in patients recovering from a recent stroke. Secondary, to evaluate the efficacy of SA4503 compared to placebo.

DETAILED DESCRIPTION:
Further study details as provided by M's Science Corporation:

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females 18 years of age or older
* Experienced a stroke from 48 to 72 hours before randomization
* A total score of >/=4 on the NIHSS, or >/=2 on the upper or lower extremity motor scores of the NIHSS
* Medically and neurologically stable within 24 hours prior to randomization

Key Exclusion Criteria:

* Patients with transient ischemic attack
* Patients with stroke in progression
* Unstable cardiac, hepatic, or renal disease, or other major medical disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 4 weeks

SECONDARY OUTCOMES:
NIHSS | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Muir, MD, Principal Investigator — Southern General Hospital, Glasgow
Locations (1):
- Southern General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Derived] Urfer R, Moebius HJ, Skoloudik D, Santamarina E, Sato W, Mita S, Muir KW; Cutamesine Stroke Recovery Study Group. Phase II trial of the Sigma-1 receptor agonist cutamesine (SA4503) for recovery enhancement after acute ischemic stroke. Stroke. 2014 Nov;45(11):3304-10. doi: 10.1161/STROKEAHA.114.005835. Epub 2014 Sep 30. PMID 25270629